CLINICAL TRIAL: NCT06452446
Title: Telehealth-based Symptom Management for Veterans Treated With Selinexor
Acronym: Selinexor
Status: Active, not recruiting | Type: Observational
Sponsor: Durham VA Medical Center (U.S. Federal Agency)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: 1749975
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma; Large-cell Lymphoma
MeSH Terms: conditions — Multiple Myeloma; Dendritic Cell Sarcoma, Interdigitating | interventions — selinexor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Selinexor — Selinexor is an oral therapy that is FDA approved for multiple myeloma and diffuse large B-cell lymphoma that have returned after prior therapy. Side effects like nausea, vomiting, and fatigue can affect how long a patient is able to continue taking Selinexor, which could mean that treatment might stop sooner.
  Other Names: Xpovio

SUMMARY:
The purpose of this study is to find out if continued monitoring of side effects from Selinexor and prescribed medication to prevent side effects helps improve symptoms, quality of life, and ability to continue the treatment longer.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate control of treatment-related and cancer-associated symptoms over the first three months of therapy with selinexor in Veterans who participate in a telehealth symptom management intervention.

The secondary objectives are:

* To describe characteristics of patients treated with selinexor.
* To describe adherence with the telehealth intervention.
* To define the type and frequency of adverse events that patients experience while taking selinexor.
* To describe the duration of selinexor therapy and evaluate adherence and dose intensity of selinexor in VA cancer patients receiving a telehealth symptom management intervention.
* To describe concomitant medication usage in patients treated with selinexor.
* To assess quality of life in patients treated with selinexor in the VA.
* To estimate progression-free survival in VA cancer patients treated with selinexor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of B-cell malignancy: either relapsed or refractory multiple myeloma or diffuse large B-cell lymphoma, meeting the FDA-approved indication for Selinexor treatment.
* Requiring therapy as assessed by the treating oncology provider.
* Prior authorization drug request for selinexor approved by VA oncology pharmacist.
* Subject age 18 years or older.
* Subject willing and able to perform video or telephone research visits.
* Subjects must be able to read and comprehend English.
* Subject must be a Veteran receiving cancer care from a VA facility affiliated with the National Teleoncology Program.
* Patients must be enrolled prior to starting Selinexor.

Exclusion Criteria:

* Any prior or current therapy with selinexor.
* Any medical, psychiatric, or cognitive issue that the principal investigator or the subject's oncologists believes would prevent participation or completion of the study.
* Individuals who are vulnerable to coercion or undue influence.
* Any individuals or populations that may temporarily or permanently require additional considerations include such as those susceptible to coercion or undue influence (e.g., patients with limited or no treatment options, socially and economically disadvantaged persons).
* Current selinexor therapy that is part of an investigational clinical trial.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrolled subjects will be Veterans with either relapsed/refractory multiple myeloma or diffuse large B-cell lymphoma who will be initiating Selinexor or Selinexor-based therapy, as recommended by treating oncologist.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | 2 years
  • VSAS: Veteran Symptom Assessment Scale (VSAS), a cancer symptom measurement tool.
Primary Outcome Measure | 2 years
  • CTCAE: Common Terminology Criteria for Adverse Events, version 5.0, an adverse event measuring tool used in clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Friedman, MD, Principal Investigator — Durham VA Medical Center
Locations (1):
- Durham VA Medical Center, Durham, North Carolina, United States